CLINICAL TRIAL: NCT01119365
Title: Bright Light as a Countermeasure for Circadian Desynchrony
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Stanford University (Other); Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Associate Professor, VA Palo Alto Health Care System
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 10165
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: Healthy controls

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator is unaware of specific sequence of light that is given to the participant until all data are analyzed.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Light (Experimental): Sequence of bright light flashes of varying durations, interflash intervals, flash lengths, flash brightness, and flash color.
  Interventions: Other: Bright light

INTERVENTIONS:
Other: Bright light — Light is administered through a custom designed mask with LED lights.

SUMMARY:
Light is the primary means by which the internal circadian clock remains aligned ("entrained") with the external world. Misalignment of this internal clock can occur during situations such as shift work and jet travel across multiple time zones (jet lag). The purpose of this study is to examine how sequences of brief flashes of light can affect entrainment of the clock.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* Normal hearing

Exclusion Criteria:

* Sleep disorder
* Extreme chronotype
* Regular smoker
* Depression
* Alcohol abuse
* Illegal drug use

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Circadian phase | 2 days
  The timing of the onset of melatonin is compared before and after a light stimulus

SECONDARY OUTCOMES:
Alertness | 1 hour
  Alertness as assessed through change in brain wave (electroencephalographic, EEG) activity, questionnaires, and objective testing is examined before and at the end of a light stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Zeitzer, PhD, Principal Investigator — Stanford University/VAPAHCS
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Background] Zeitzer JM, Dijk DJ, Kronauer R, Brown E, Czeisler C. Sensitivity of the human circadian pacemaker to nocturnal light: melatonin phase resetting and suppression. J Physiol. 2000 Aug 1;526 Pt 3(Pt 3):695-702. doi: 10.1111/j.1469-7793.2000.00695.x. PMID 10922269
- [Background] Cajochen C, Zeitzer JM, Czeisler CA, Dijk DJ. Dose-response relationship for light intensity and ocular and electroencephalographic correlates of human alertness. Behav Brain Res. 2000 Oct;115(1):75-83. doi: 10.1016/s0166-4328(00)00236-9. PMID 10996410
- [Background] Zeitzer JM, Khalsa SB, Boivin DB, Duffy JF, Shanahan TL, Kronauer RE, Czeisler CA. Temporal dynamics of late-night photic stimulation of the human circadian timing system. Am J Physiol Regul Integr Comp Physiol. 2005 Sep;289(3):R839-44. doi: 10.1152/ajpregu.00232.2005. Epub 2005 May 12. PMID 15890792
- [Result] Zeitzer JM, Ruby NF, Fisicaro RA, Heller HC. Response of the human circadian system to millisecond flashes of light. PLoS One. 2011;6(7):e22078. doi: 10.1371/journal.pone.0022078. Epub 2011 Jul 8. PMID 21760955
- [Result] Zeitzer JM, Fisicaro RA, Ruby NF, Heller HC. Millisecond flashes of light phase delay the human circadian clock during sleep. J Biol Rhythms. 2014 Oct;29(5):370-6. doi: 10.1177/0748730414546532. Epub 2014 Sep 16. PMID 25227334
- [Result] Najjar RP, Zeitzer JM. Temporal integration of light flashes by the human circadian system. J Clin Invest. 2016 Mar 1;126(3):938-47. doi: 10.1172/JCI82306. Epub 2016 Feb 8. PMID 26854928
- [Result] Joyce DS, Spitschan M, Zeitzer JM. Duration invariance and intensity dependence of the human circadian system phase shifting response to brief light flashes. Proc Biol Sci. 2022 Mar 9;289(1970):20211943. doi: 10.1098/rspb.2021.1943. Epub 2022 Mar 9. PMID 35259981